CLINICAL TRIAL: NCT04368507
Title: A Phase 1b/2a Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of YYB101, Hepatocyte Growth Factor (HGF)-Neutralizing Humanized Monoclonal Antibody (Mab) in Combination With Irinotecan in Metastatic or Recurrent Colorectal Cancer Patients
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of YYB101 With Irinotecan, Patients Who Are Metastatic or Recurrent Colorectal Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CellabMED (Industry)
Collaborators: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV110501-201
Record Dates: First submitted 2019-11-24; First posted 2020-04-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Recurrent
MeSH Terms: interventions — monoclonal antibody YYB-101

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YYB101+Irinotecan (Experimental): 1. b (Dose level 0 cohort): YYB101 20mg/kg, Irinotecan 150 mg/m2 of each dose level, IV infusion on Day 1, Day15, and followed by every 2 weeks
  2. a Stage 1: YYB101 RP2D, Irinotecan 150 mg/m2 of each dose level, IV infusion on Day 1, Day15, and followed by every 2 weeks
  Interventions: Drug: YYB101

INTERVENTIONS:
Drug: YYB101 — 1. b (Dose level 0 cohort): YYB101 20mg/kg, Irinotecan 150 mg/m2 of each dose level, IV infusion on Day 1, Day15, and followed by every 2 weeks until disease progression or unacceptable toxicity
  2. a Stage 1: YYB101 RP2D, Irinotecan 150 mg/m2 of each dose level, IV infusion on Day 1, Day15, and followed by every 2 weeks until disease progression or unacceptable toxicity

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and antitumor activity of YYB101 with Irinotecan, patients who are metastatic or recurrent Colorectal Cancer Patients.

DETAILED DESCRIPTION:
Metastatic or recurrent colorectal cancer patients will be enrolled to evaluate the safety, tolerability, pharmacokinetics, and efficacy of YYB101 in combination with irinotecan. In Phase 1b, YYB101 20 mg/kg in combination with irinotecan 150 mg/m2 will be administered as a dose level 0, and the safety and pharmacokinetic assessments will be performed based on the DLT after a 4-week treatment period. If no DLT occurs during the 4-week observation period, dosing will be continued every 2 weeks until progressive disease (PD) or unacceptable toxicity occurs. After completion of Phase 1b, the SRC will determine the RP2D of YYB101 and irinotecan, and Phase 2a will be initiated. Stage 2 will proceed when unconfirmed response is observed in one or more subjects out of 10 subjects evaluable for tumor in Phase 2a Stage 1 which includes the RP2D dose cohort in Phase 1b.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 19 years
2. Patients with histologically confirmed metastatic or recurrent colorectal cancer

   * Patients who progressed after standard anticancer treatment including existing fluoropyrimidine, oxaliplatin, and irinotecan
   * Patients who received anticancer treatment including irinotecan for at least 6 weeks, with progression confirmed radiologically while on anticancer treatment or within 6 months (24 weeks) after completion of anticancer treatment
   * Adjuvant therapy is acknowledged as an anticancer therapy, if PD is confirmed within 6 months (24 weeks) after the last dose
   * Patients who are unable to undergo radical resection 3) Patients with Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 4) Patients with life expectancy of at least 12 weeks 5) Patients with confirmed adequate hematologic, renal and hepatic function based on the following criteria:
   * ANC ≥ 1,500/μL (without granulocyte colony-stimulating factor (G-CSF) administration within 2 weeks prior to baseline)
   * Platelet ≥ 100,000/μL (without transfusion within 2 weeks prior to baseline)
   * Hemoglobin ≥ 9 g/dL (without transfusion within 4 weeks prior to baseline)
   * Serum creatinine ≤ 1.5 mg/dL or estimated glomerular filtration rate (eGFR) (or GFR) ≥ 60 mL/min/1.73 m2
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 X upper limit of normal (ULN) (AST and ALT ≤ 5 X ULN for subjects with confirmed hepatic metastases)
   * Total bilirubin ≤ 1.5 X ULN
   * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN
   * Urine protein to creatinine ratio (UPC) < 1.0 0 (g/g)a a UPC will be conducted only when urine dipstick protein level is ≥ 1 positive (+).

6. Patients with a measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 7. Patients who voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Patients with hematologic malignancy including lymphoma
2. Patients who received chemotherapy, biological therapy, immunotherapy (including immune checkpoint inhibitors), or radiotherapy within 4 weeks prior to baseline for the treatment of metastatic or recurrent colorectal cancer (Participation is not allowed if nitrosoureas or mitomycin is administered within 6 weeks prior to baseline or if biological target antibody is administered within 8 weeks prior to baseline)
3. Patients with a history of primary malignancy other than colorectal cancer. However, the patients are permitted to participate if:

   * They have not received any treatment for the tumor or are disease-free for at least 5 years (For papillary carcinoma of thyroid, participation in the study is allowed even if it has not been more than 5 years after radical resection.)
   * At least 1 year has passed since complete resection of basal/squamous cell carcinoma of the skin or successful treatment of cervical carcinoma in situ
4. Patients with symptomatic central nervous system metastases (except for patients who have discontinued systemic corticosteroid treatment at least 4 weeks prior to baseline and are neurologically stable for at least 4 weeks)
5. Patients with the following medical or surgical/procedural history

   * Deep vein thrombosis (DVT) or pulmonary embolism (PE) within 1 year prior to baseline
   * History of infection with cytomegalovirus (CMV) or Epstein-Barr virus (EBV) within 6 months (24 weeks) prior to baseline
   * History of acute coronary syndrome (unstable angina or myocardial infarction) within 6 months (24 weeks) prior to baseline
   * Serious cerebrovascular disease such as stroke within 6 months (24 weeks) prior to baseline
   * Major surgery that requires general anesthesia or a ventilation assist within 4 weeks prior to baseline (within 2 weeks for video-assisted thoracoscopic surgery [VATS] or open-and-closed [ONC] surgery)
6. Patients with any of the following diseases:

   * New York Heart Association (NYHA) class III or IV heart failure
   * Uncontrolled hypertension (SBP > 160 mmHg or DBP > 90 mmHg despite drug treatments)
   * Clinically significant cardiovascular abnormalities as determined by the investigator (e.g., left ventricular ejection fraction [LVEF] < 50%, clinically significant abnormal cardiac wall or myocardial injury, or uncontrolled cardiac arrhythmias)
   * Known positive human immunodeficiency virus (HIV)
   * Severe infection requiring systemic antibiotics, antivirals, etc. or other uncontrolled acute active infectious diseases
   * Chronic inflammatory bowel disease
   * Severe enteroplegia or ileus requiring intervention
   * Pneumonitis or pulmonary fibrosis
   * Large amount of ascites or pleural fluid
   * Diarrhea (watery stool)
7. Patients requiring continued treatment with systemic corticosteroids
8. Patients on antithrombotic agents (patients on low dose aspirin of < 325 mg for inhibition of platelet aggregation is allowed to participate) or with a predisposition to bleeding, large amount of hemoptysis, gastrointestinal hemorrhage or peptic ulcers
9. Patients with a history of severe drug hypersensitivity or hypersensitivity to class of drugs similar to the study drug/concurrent medications
10. Pregnant or breast-feeding women
11. Women of childbearing potential and men who are unwilling to remain abstinent or use appropriate methods of contraception during the study and for at least 5 months (20 weeks) following the end of treatment
12. Patients who received other investigational product or used any investigational device within 4 weeks prior to baseline
13. Patients considered ineligible to participate in the clinical study according to the investigator's judgement for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
1b (Dose level 0) cohort: Safety, Tolerability of YYB101 by DLTs and MTD | 28 days
  DLTs and MTD
2a cohort: Safety, Tolerability of YYB101 by ORR | By 12 months after enrollment of the last subject
  ORR

SECONDARY OUTCOMES:
1b (Dose level 0) cohort | By 12 months after enrollment of the last subject
  Safety and tolerability (MTD/RP2D based by DLT, Incidence of AEs that result in discontinuation and dose reduction of YYB101, Clinical laboratory abnormalities that result in discontinuation and dose reduction of YYB101, Vital sign that result in discontinuation and dose reduction of YYB101, Anti-YYB101 antibody that result in discontinuation and dose reduction of YYB101)
1b (Dose level 0) cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Area under the plasma concentration versus time curve (AUC)
1b (Dose level 0) cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Peak Plasma Concentration (Cmax)
1b (Dose level 0) cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Serum HGF Concentration profile
1b (Dose level 0) cohort | By 12 months after enrollment of the last subject
  Antitumor activity of YYB101 and Irinotecan (Tumor response result evaluted by RECIST version 1.1)
2a cohort | By 12 months after enrollment of the last subject
  Progression-free survival (PFS) will be measured using RECIST version 1.1
2a cohort | By 12 months after enrollment of the last subject
  Disease Control Rate (DCR) will be measured using RECIST version 1.1
2a cohort | By 12 months after enrollment of the last subject
  Duration Of Response (DOR) will be measured using RECIST version 1.1
2a cohort | By 12 months after enrollment of the last subject
  Overall Survival (OS) will be measured using RECIST version 1.1
2a cohort | By 12 months after enrollment of the last subject
  Safety profile (Incidence of AEs that result in discontinuation and dose reduction of YYB101, Clinical laboratory abnormalities that result in discontinuation and dose reduction of YYB101, Vital sign that result in discontinuation and dose reduction of YYB101, Anti-YYB101 antibody that result in discontinuation and dose reduction of YYB101)
2a cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Area under the plasma concentration versus time curve (AUC)
2a cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Peak Plasma Concentration (Cmax)
2a cohort | By 12 months after enrollment of the last subject
  Pharmacokinetics: Serum HGF Concentration profile [only stage 1 subject]

CONTACTS AND LOCATIONS:
Overall Officials: Hoonkyo Kim, Ph.D, Study Director — National OncoVenture/National Cancer Center; Garam Im, Study Director — National OncoVenture/National Cancer Center
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Seoul, Goyang-si, Gyeonggi-do
  - Seoul ST. Mary's Hospital, Seoul, Seocho-gu

IPD SHARING:
Plan to Share IPD: Undecided